CLINICAL TRIAL: NCT00065130
Title: Safety and Efficacy of Insulin Aspart vs. Regular Human Insulin in Basal/Bolus Therapy for Patients With Gestational Diabetes
Brief Title: Safety and Efficacy of Insulin Aspart vs. Regular Human Insulin in Gestational Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANA-2067
Record Dates: First submitted 2003-07-17; First posted 2003-07-18 (Estimated); Last update posted 2016-12-22 (Estimated); Status verified 2016-12

CONDITIONS: Diabetes; Gestational Diabetes
MeSH Terms: conditions — Diabetes Mellitus; Diabetes, Gestational | interventions — Insulin; Insulin, Isophane; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: human insulin
Drug: insulin NPH
Drug: insulin aspart

SUMMARY:
This trial is conducted in the United States of America (USA). The purpose of this study is to test whether NovoLog (insulin aspart) is a safe and at least as effective alternative to regular human insulin for the control of blood glucose after meals in women who develop diabetes during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects older than 35 years old will be considered
* Gestational diabetes mellitus

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2000-04; Primary Completion 2003-12 (Actual); Study Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
Postprandial glycemic control

SECONDARY OUTCOMES:
HbA1c (glycosylated haemoglobin A1c)
Postprandial endogenous insulin secretory response
Hypoglycemic episodes
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Santa Barbara, California, United States

REFERENCES:
- [Result] Pettitt DJ, Ospina P, Kolaczynski JW, Jovanovic L. Comparison of an insulin analog, insulin aspart, and regular human insulin with no insulin in gestational diabetes mellitus. Diabetes Care. 2003 Jan;26(1):183-6. doi: 10.2337/diacare.26.1.183. PMID 12502678
- [Result] Pettitt DJ, Ospina P, Howard C, Zisser H, Jovanovic L. Efficacy, safety and lack of immunogenicity of insulin aspart compared with regular human insulin for women with gestational diabetes mellitus. Diabet Med. 2007 Oct;24(10):1129-35. doi: 10.1111/j.1464-5491.2007.02247.x. PMID 17888133
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com